CLINICAL TRIAL: NCT00898560
Title: Effect of Repeated Administration of Eslicarbazepine Acetate (BIA 2-093) 800mg Once-daily on the Pharmacokinetics of a Combined Oral Contraceptive in Healthy Female Subjects
Brief Title: Effect of Repeat Administration of Eslicarbazepine Acetate on the Pharmacokinetics of a Combined Oral Contraceptive
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-128
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Partial Epilepsy
Keywords: Partial; Epilepsy; Eslicarbazepine acetate; Combined oral contraceptive; Pharmacokinetics; Tolerability
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Microginon® (Other): A single oral dose of a combined oral contraceptive containing 30ug ethinyloestradiol and 150ug levonorgestrel (Microginon ®).
  Interventions: Drug: Microginon®
- ESL and Microginon® (Experimental): 15-day treatment with ESL 800 mg once daily, with co administration of a single oral dose of Microginin® on Day 14 of the relevant dosing period, to assess impact of ESL on pharmacokinetics of the combined oral contraceptive.
  Interventions: Drug: eslicarbazepine acetate and Microginon®

INTERVENTIONS:
Drug: eslicarbazepine acetate and Microginon® — eslicarbazepine acetate: once-daily oral dose of 800 mg on days 1- 15 of treatment period.
  Microginon®: single oral dose on day 14 of treatment period
  Other Names: ESL; BIA 2-093
  Arms: ESL and Microginon®
Drug: Microginon® — Single oral dose of Microginon® (30ug ethinyloestradiol and 150ug levonorgestrel)
  Arms: Microginon®

SUMMARY:
The purpose of this study is to investigate whether multiple-dose administration of eslicarbazepine acetate (ESL, BIA 2-093) 800 mg once-daily (QD) affects the pharmacokinetics and tolerability of the components of a combined oral contraceptive (ethinyloestradiol and levonorgestrel).

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal female subjects
* Age 18-40 years, inclusive
* Body mass index (BMI) 19-30 kg/m2, inclusive
* Healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG
* Negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening
* Negative urine pregnancy test at screening and admission to each treatment period.
* Using one of the following methods of contraception: double barrier or intrauterine device

Exclusion Criteria:

* Subjects who have any contra-indication to the use of oral contraceptives
* History or presence of clinically relevant diseases, disorders or surgical history
* History of alcoholism or drug abuse
* Have used medicines within two weeks of admission to first period that may affect the safety or other study assessments, in the investigator's opinion

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Vaz-da-Silva, Principal Investigator — Bial Portela
Locations (1):
- Human Pharmacology Unit (UFH), Section of Clinical Research (SIC), Department of Research & Development (DID), BIAL - Portela & Cª, SA, S. Mamede do Coronado, Porto, Portugal

RESULTS

PARTICIPANT FLOW:
Groups:
- ESL and Microginon®: 15-day treatment with ESL 800 mg once daily, with co administration of a single oral dose of Microginin® on Day 14 of the relevant dosing period, to assess impact of ESL on pharmacokinetics of the combined oral contraceptive.
  eslicarbazepine acetate and Microginon®: eslicarbazepine acetate: once-daily oral dose of 800 mg on days 1- 15 of treatment period.
  Microginon®: single oral dose on day 14 of treatment period
Period: Overall Study
Arm/Group | ESL and Microginon®
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | ESL and Microginon®
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Concentration
Description: To investigate whether multiple-dose administration of eslicarbazepine acetate (ESL, BIA 2-093) 800 mg once-daily (QD) affects the pharmacokinetics of the components of a combined oral contraceptive (ethinyloestradiol and levonorgestrel).
Time Frame: 15-day
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Microginon® | ESL and Microginon®
Number analyzed (Participants) | 19 | 19
pg/mL
  Cmax (ethinyloestradiol) | 82.4 (23.4) | 75.0 (26.8)
  Cmax (levonogestrel) | 4170 (1720) | 4340 (1530)

2. Secondary Outcome: AUC0-t - Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Sampling Time at Which Concentrations Were at or Above the Limit of Quantification
Description: as for outcome 1
Time Frame: 15-day
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Microginon® | ESL and Microginon®
Number analyzed (Participants) | 19 | 19
ng.h/mL
  AUC0-t (ethinyloestradiol) | 0.665 (0.195) | 0.453 (0.167)
  AUC0-t (levonogestrel) | 37.4 (19.1) | 32.0 (12.9)

3. Secondary Outcome: AUC0-∞ - Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity
Description: as for outcome 1
Time Frame: 15-day
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Microginon® | ESL and Microginon®
Number analyzed (Participants) | 19 | 19
ng.h/mL
  AUC0-∞ (ethinyloestradiol) | 0.768 (0.223) | 0.533 (0.181)
  AUC0-∞ (levonorgestrel) | 52.1 (22.1) | 43.1 (13.3)

ADVERSE EVENTS:
Arm/Group | ESL and Microginon® | Microginon®
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 18/20 | 8/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ESL and Microginon® (N=20) | Microginon® (N=20)
Xerophthalmia (Eye disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dry throat (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 0
Paraesthesia oral (Gastrointestinal disorders) | 5 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Vessel puncture site haematoma (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 1
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Diplopia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 5 | 0
Headache (Nervous system disorders) | 6 | 2
Somnolence (Nervous system disorders) | 8 | 2
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Libido increased (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cheilitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Sexual activity increased (Social circumstances) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No